CLINICAL TRIAL: NCT02947347
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With Rituximab Versus Placebo in Combination With Rituximab in Treatment Naïve Subjects With Follicular Lymphoma (PERSPECTIVE)
Brief Title: Study of Ibrutinib and Rituximab in Treatment Naïve Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCYC-1141-CA; 2016-003202-14 (EudraCT Number)
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (Arm A) ibrutinib + rituximab (Experimental): Participants will receive 560mg of ibrutinib and rituximab 375mg/m^2 weekly x4 with maintenance.
  Interventions: Drug: ibrutinib; Drug: rituximab
- (Arm B) placebo + rituximab (Placebo Comparator): Participants will receive placebo and rituximab 375mg/m^2 weekly x4 with maintenance.
  Interventions: Drug: placebo to match ibrutinib; Drug: rituximab

INTERVENTIONS:
Drug: ibrutinib — ibrutinib 560mg administered orally
  Other Names: Imbruvica
  Arms: (Arm A) ibrutinib + rituximab
Drug: placebo to match ibrutinib — placebo capsules to match ibrutinib administered orally
  Arms: (Arm B) placebo + rituximab
Drug: rituximab — rituximab 375mg/m^2 IV

SUMMARY:
The purpose of this study is to evaluate whether the addition of ibrutinib will result in prolongation of progression-free survival (PFS) when compared with rituximab alone in treatment naïve participants with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma CD20+ (Grade 1, 2 or 3a) Ann Arbor Stage II, III or IV disease.
* Measurable disease
* Subjects 70 years of age or older; OR subjects 60-69 years of age who have one or more comorbidities.
* Meets one or more Groupe d'Etude des Lymphomes Folliculaire (GELF) criteria.
* Adequate hematologic function within protocol-defined parameters.
* Adequate hepatic and renal function within protocol-defined parameters.
* ECOG performance status score of 0-2.

Exclusion Criteria:

* Transformed lymphoma
* Prior treatment for follicular lymphoma.
* Central nervous system lymphoma or leptomeningeal disease.
* Currently active, clinically significant cardiovascular disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Progression-Free Survival (PFS) | 2-5 years
  PFS, is assessed by the investigator, will be analyzed in the intent to treat (ITT) population, comparing the 2 treatment arms (Arm A and Arm B).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 2-5 years
  ORR of the two treatment arms will be compared using the Cochran-Mantel-Haenszel (CMH) chi-square test, stratified by the randomization stratification factors, under the hierarchical procedure.
Overall Survival | 2-5 years
  Overall survival is defined as the interval between the date of randomization and the date of the participant's death from any cause.
Infusion-Related Reaction Rate | 2-5 years
  Infusion-related reaction rate Arm A vs. Arm B.
Duration of Response (DOR) as Assessed by Investigator | 2-5 years
  DOR is defined as the time from the date of the participant's documented disease progression or death due to the disease, whichever occurs first.
Number of Participants with Adverse Events (AE) | 2-5 years
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (128):
- United States (25):
  - Southern Cancer Center, Mobile, Alabama
  - City of Hope, Duarte, California
  - Sansum Clinic, Santa Barbara, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Helen F. Graham Cancer Center and Research Institute, Newark, Delaware
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Affiliates, Ocala, Florida
  - SCRI Florida Cancer Specialists North, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - OHSU Knight Cancer Institute Beaverton Clinic, Beaverton, Oregon
  - Greenville Health System, Greenville, South Carolina
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
  - Texas Oncology (Medical City), Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - SCRI The Center For Cancer and Blood Disorders, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology (Tyler), Tyler, Texas
  - Oncology and Hematology Associates of Southwest Virginia (Blacksburg), Blacksburg, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - W VA University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Mater Misericordiae Health Services, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre Clayton Campus, Clayton, Victoria
  - Andrew Love Cancer Center, Geelong, Victoria
- Austria (2):
  - Universitätsklinikum Innsbruck, Innsbruck, Tyrol
  - Uniklinikum Salzburg, Salzburg
- Belgium (7):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - ZNA Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge Oostende AV, Bruges
  - UZ Gent, Ghent
  - CHU de Liège, Liège
  - AZ Nikolaas, Sint-Niklaas
  - Gasthuis Zusters Antwerpen, Wilrijk
- Canada (3):
  - Moncton Hospital, Moncton, New Brunswick
  - CHUM Notre Dame Hospital, Montreal, Quebec
  - CIUSSS-de-l'Est-de-l'Île-de-Montréal, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
- France (6):
  - Centre Hospitalier de Valence, Valence, Drôme
  - CHRU de Poitiers La Miletrie, Poitiers, Vienne
  - CHU de Limoges Hôpital Dupuytren, Limoges
  - CHU Bordeaux, Pessac
  - Centre Hospitalier de Perigueux, Périgueux
  - Hôpital Civil, Strasbourg
- Greece (3):
  - University General Hospital of Patras, Pátrai, Achaïa
  - Laiko General Hospital of Athens, Athens, Attica
  - University General Hospital of Larissa, Larissa
- Hungary (5):
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Országos Onkológiai Intézet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Pécsi Tudományegyetem, Pécs
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Bnei Zion Medical Center, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Assuta Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Ẕerifin
- Italy (14):
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda ospedaliera Universiataria Senese, Siena, Tuscany
  - Centro Di Riferimento Oncologico, Aviano
  - Azienda Sanitaria Ospedaliera S. Croce e Carle, Cuneo
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST, Meldola
  - San Raffaele Scientific Institute, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Farmacia Polo Ematologico Policlinico Umberto I, Roma
  - Policlinico Universitario Campus Biomedico di Roma, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Netherlands (4):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Leids Universitair Medisch Centrum, Leiden
  - ETZ-Elisabeth, Tilburg
- Poland (5):
  - Centrum Onkologii Ziemi Lubelskiej, Lublin, Lublin Voivodeship
  - Copernicus PL Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
  - Malopolskie Centrum Medyczne, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Portugal (4):
  - Unidade Local de Saúde de Matosinhos SA, Matosinhos Municipality
  - Centro Hospitalar de São João, E.P.E., Porto
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
- Russia (5):
  - Regional Clinical Hospital, Krasnoyarsk
  - Russian Oncology Research Center n a N N Blokhin, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - City Hospital #31, Saint Petersburg
  - North-West Federal Medical Research Center n.a. V.A. Almazov, Saint Petersburg
- Spain (11):
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Virgen de Valme, Seville, Sevilla
  - Hospital del Mar, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Vall dHebron, Barcelona
  - ICO L'Hospitalet, Barcelona
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Taiwan (5):
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chi Mei Medical Center, Liouying, Liuying
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (7):
  - Gazi Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ege Universitesi Tip Fakultesi Hastanesi, Bornova
  - Mersin Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Arastirma ve Uygulama Hastanesi, Kocaeli
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Namik Kemal Universitesi Tip Fakultesi Hastanesi, Tekirdağ
- United Kingdom (7):
  - Royal Cornwall Hospital - Hospital Treliske, Tururo, Cornwall
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Addenbrooke's Hospital, Cambridge
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Barts and The London NHS Trust, London
  - Derriford Hospital, Plymouth
  - Royal Berkshire Hospital NHS Foundation Trust, Reading